CLINICAL TRIAL: NCT07021105
Title: COMPARISON OF ERECTOR SPINAE PLANE BLOCK, QUADRATUS LUMBORUM BLOCK, AND TRANSVERSUS ABDOMINIS PLANE BLOCK IN POSTOPERATIVE PAIN MANAGEMENT IN GYNECOLOGICAL ABDOMINAL SURGERIES
Brief Title: COMPARISON OF PLAIN BLOCKS FOR POSTOPERATIVE PAIN MANAGEMENT IN GYNECOLOGICAL ABDOMINAL SURGERIES
Acronym: ESP QLB TAP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Hakki Unlugenc, Prof Dr, Cukurova University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Decision No. 145
Record Dates: First submitted 2025-05-21; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Surgery With General Anesthesia; Gynecologic Surgical Procedures; Plane Block; Postoperative Pain Management
Keywords: Gynecologic surgery; Transversus abdominis plane block; Erector spinae plaen block; Quadratus lumborum block; morphine consumption

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned into four groups using a computer-generated randomization method. According to group allocation, patients will receive the following interventions before extubation under ultrasound (US) guidance except control group.
  Group E (n=20): Bilateral erector spinae plane (ESP) block Group Q (n=20): Bilateral quadratus lumborum block (QLB) Group T (n=20): Bilateral transversus abdominis plane (TAP) block Group C (Control group, n=20): No block will be applied
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group E (Active Comparator): Group ESP & QLB, TAP, Control
  Interventions: Procedure: QLB plane block; Procedure: TAP Block; Other: No intervention
- Group Q (Active Comparator): Group QLB & ESP, TAP, Control
  Interventions: Procedure: ESP Plane block; Procedure: TAP Block; Other: No intervention
- Group T (Active Comparator): Group T & ESP, QLB, Control
  Interventions: Procedure: ESP Plane block; Procedure: QLB plane block; Other: No intervention
- Group C (No Intervention): Group C & ESP, QLB, TAP

INTERVENTIONS:
Procedure: ESP Plane block — Group E (n=20): Bilateral erector spinae plane (ESP) block will be performed with 40 ml of 0.25% bupivacaine (20 ml on each side) at the T12 level, approximately 3-4 cm laterally from the midline, in the neurofascial plane between the transverse processes and the erector spinae muscle.
  Arms: Group Q; Group T
Procedure: QLB plane block — Group Q (n=20): Bilateral quadratus lumborum block (QLB) will be performed with 40 ml of 0.25% bupivacaine (20 ml on each side), placed between the psoas major and quadratus lumborum muscles under US guidance, between the iliac crest and the 12th rib.
  Arms: Group E; Group T
Procedure: TAP Block — Group T (n=20): Bilateral transversus abdominis plane (TAP) block will be performed with 40 ml of 0.25% bupivacaine (20 ml on each side) in the neurofascial plane between the internal oblique and transversus abdominis muscles.
  Arms: Group E; Group Q
Other: No intervention — Group C (Control group, n=20): No block will be applied, only the standard intravenous patient-controlled analgesia (PCA) protocol will be used.
  Arms: Group E; Group Q; Group T

SUMMARY:
This study compares the effects of transversus abdominis plane (TAP) block, quadratus lumborum block (QLB), and erector spinae plane block (ESP) on postoperative morphine consumption, pain scores, patient satisfaction, and side effects in patients undergoing gynecological abdominal laparotomy surgeries.

DETAILED DESCRIPTION:
Patients will be randomly assigned into four groups using a computer-generated randomization method. According to group allocation, patients will receive the following interventions before extubation under ultrasound (US) guidance except control group:

Group E (n=20): Bilateral erector spinae plane (ESP) block will be performed with 40 ml of 0.25% bupivacaine (20 ml on each side) at the T12 level, approximately 3-4 cm laterally from the midline, in the neurofascial plane between the transverse processes and the erector spinae muscle.

Group Q (n=20): Bilateral quadratus lumborum block (QLB) will be performed with 40 ml of 0.25% bupivacaine (20 ml on each side), placed between the psoas major and quadratus lumborum muscles under US guidance, between the iliac crest and the 12th rib.

Group T (n=20): Bilateral transversus abdominis plane (TAP) block will be performed with 40 ml of 0.25% bupivacaine (20 ml on each side) in the neurofascial plane between the internal oblique and transversus abdominis muscles.

Group C (Control group, n=20): No block will be applied, only the standard intravenous patient-controlled analgesia (PCA) protocol will be used.

The primary aim of this study is to assess the morphine consumption in the postoperative period, while secondary aims include pain score, patient satisfaction, the need for rescue analgesia and side effects

ELIGIBILITY:
Inclusion Criteria:

aged between 18 and 69 years, with ASA 1-2 score scheduled to undergo major gynecological abdominal surgery

Exclusion Criteria:

ASA score 3 or above, patients younger than 18 or older than 69 years, patients with bleeding disorders or using anticoagulants, patients with a body mass index over 40, patients with known allergies to any drugs used in the study, and patients who could not or did not wish to use Patient-Controlled Analgesia (PCA) device

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 80 patients aged between 18 and 69 years, with ASA 1-2 score (mild anemia, hypertension, diabetes, obesity, etc.), who were scheduled to undergo major gynecological abdominal surgery
Enrollment: 80 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-08-11 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
morphine consumption in the postoperative period | For postoperative 24 hours
  Thus the primary aim of this study was to assess the morphine consumption in the postoperative period

SECONDARY OUTCOMES:
pain score (VAS=0-10), patient satisfaction (0-10), the need for rescue analgesia (mg) and side effects | For postoperative 24 hours
  Secondary outcomes included pain score (VAS=0-10), patient satisfaction (0-10), the need for rescue analgesia (mg) and side effects

CONTACTS AND LOCATIONS:
Overall Officials: Hakkı Ünlügenç, Professör, Study Director — Cukurova University
Locations (1):
- Cukurova University, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Considering but not decided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/